CLINICAL TRIAL: NCT02972567
Title: Evaluation of the Effect of a Lactobacillus Reuteri Strain on Markers of Inflammation, Cardiovascular Risk and Fatty Liver Disease in Obese Subjects With Insulin Resistance
Brief Title: Evaluation of the Effects of a L.Reuteri Strain on Markers of Inflammation, Cardiovascular Risk and Fatty Liver Disease
Acronym: PROSIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Collaborators: Universidad de Granada (Other); Complejo Hospitalario de Jaen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P3600
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Metabolic Syndrome X
Keywords: probiotics; metabolic syndrome; non-alcoholic fatty liver disease
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus strain
  Interventions: Dietary Supplement: Lactobacillus spp
- Control (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Lactobacillus spp — 9 log10 cfu/capsule. 1 capsule/day for 12 weeks
  Arms: Probiotic
Dietary Supplement: Control — Maltodextrin
  Arms: Control

SUMMARY:
The purpose of this study is the evaluation of the effects in obese patients with metabolic syndrome on the composition of the intestinal microbiota, markers of the syndrome (hypertension, dyslipidemia, inflammation biomarkers, risk cardiovascular and hepatic steatosis) and other possible metabolites involved.

DETAILED DESCRIPTION:
Randomized double blind crossover placebo controlled intervention study

The proposed study will be conducted by members of the Endocrinology and Nutrition Services (ENCHJ), and Gastroenterology (ADCHJ), of the Hospital of Jaen and members of the Department of Biochemistry and Molecular Biology II of the University of Granada (UGR) and members of Microbiology Department of the University Hospital San Cecilio of Granada (MHUSC).

The selection, clinical and anthropometric control, general biochemical parameters and the determination of hepatic steatosis by ultrasound will be performed by members of ENCHJ.

The determination of the composition of the intestinal microbiota will be carried out by members of the UGR together with members form the MHUSC. Inflammation and steatosis biomarkers as well as metabolic profile will be performed by members of the UGR.

The study will be conducted according to the Helsinki Rules and will be previously approved by the Ethics Committee of Research of Jaen. The study will follow the rules of international, national and regional research The biological samples will be managed and processed in accordance with the research protocols by the Biobanco del Sistema Sanitario Público de Andalucía. At the end of the project, samples will be stored within the framework of Biobank from Public Health Organization of Andalusia .

The present study involves access and use of information confidential, so all the data will be treated anonymously.

• Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.

Based on the range and median value on plasma lipopolysaccharide (LPS), and assuming a power of 90% and a type error alpha of 5%, the minimum number of subjects was 32. To avoid possible bias caused by gender and taking into account the withdrawal, will be recruited 60 subjects.

The missing data will be considered as unavailable data.

All statistical analyses will be performed using the statistical package SPSS (Statistical Product and Service Solutions). Normally distributed data will be expressed as the mean and standard error of the mean, whereas median and ranges will be used for data not normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of insulin resistance syndrome, according to Criteria of the International Diabetes Federation (IDF)
* BMI>30 kg/m2 or Waist Circumference ≥ 94cm (men) WC≥ 80cm (women)
* Serum Triglycerides ≥ 150 mg/dl
* HDLcholesterol < 40 mg/dl (1,03 mmol/l) in men and < 50 mg/dl (1,29 mmol/l) in women
* Systolic blood pressure ≥ 130 mmHg or diastolic ≥ 85 mmHg
* Glucose ≥ 100 mg/dl (5,6 mmol/l) (not previous diagnostic of diabetes II)

Exclusion Criteria:

* Patients with renal or hepatic impairment
* Patients with a diagnosis of diabetes
* Patients with diseases that condition immunosuppression
* Patients presenting positive serologies for liver viruses
* Being on antihypertensive treatment: beta-blockers, Angiotensin 2 receptor antagonists (ARA 2), enzyme inhibitors, Angiotensin converting enzyme (ACE) inhibitors.
* Patients receiving lipid-lowering and / or hypoglycemic agents
* Patients on treatment with drugs that increase hepatic enzymes,such as Amiodarone, perhexiline, maleate and 4,4'-diethylaminoethoxyhexestrol, synthetic estrogens, Tamoxifen, corticosteroids, acetylsalicylic acid, Valproic acid, tetracyclines, viral agents (zidovudine, zalcitabine, didanosine), among others.
* Exhibiting high values of C-reactive protein (CRP) or Sedimentation (ESR)
* Consuming alcohol in quantities greater than 40 g / d or other hepatotoxic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from basal plasma lipopolysaccharide (LPS) at 12 weeks | Basal (T0), 12 weeks

SECONDARY OUTCOMES:
Change from basal Blood pressure at 12 weeks | Basal (T0), 12 weeks
Change from basal HOMA ( homeostatic model assessment ) index at 12 weeks | Basal (T0), 12 weeks
Change from basal plasma cholesterol level (total, LDL and HDL) at 12 weeks | Basal (T0), 12 weeks
Change from basal plasma Inflammatory markers (sVCAM, sICAM, myeloperoxidase selectin, adiponectin, plasminogen activator inhibitor and resistin, and interleukines Il-6, Il-8, tumor necrosis factor, HGF, leptin and Multicopper oxidase-1) at 12 weeks | Basal (T0), 12 weeks
Change from basal Hepatic Steatosis markers (arginase, prolidase and RBP-4(Retinol binding protein-4)) at 12 weeks | Basal (T0), 12 weeks
Changes from basal fecal microbiota at 12 weeks | Basal (T0), 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gil Ángel, Prof. Ph.D, Study Director — University of Granada (Spain)
Locations (1):
- Complejo Hospitalario Universitario de Jaen, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Result] Backhed F, Manchester JK, Semenkovich CF, Gordon JI. Mechanisms underlying the resistance to diet-induced obesity in germ-free mice. Proc Natl Acad Sci U S A. 2007 Jan 16;104(3):979-84. doi: 10.1073/pnas.0605374104. Epub 2007 Jan 8. PMID 17210919
- [Result] Bermudez-Brito M, Munoz-Quezada S, Gomez-Llorente C, Matencio E, Bernal MJ, Romero F, Gil A. Human intestinal dendritic cells decrease cytokine release against Salmonella infection in the presence of Lactobacillus paracasei upon TLR activation. PLoS One. 2012;7(8):e43197. doi: 10.1371/journal.pone.0043197. Epub 2012 Aug 14. PMID 22905233
- [Derived] Tenorio-Jimenez C, Martinez-Ramirez MJ, Tercero-Lozano M, Arraiza-Irigoyen C, Del Castillo-Codes I, Olza J, Plaza-Diaz J, Fontana L, Migueles JH, Olivares M, Gil A, Gomez-Llorente C. Evaluation of the effect of Lactobacillus reuteri V3401 on biomarkers of inflammation, cardiovascular risk and liver steatosis in obese adults with metabolic syndrome: a randomized clinical trial (PROSIR). BMC Complement Altern Med. 2018 Nov 20;18(1):306. doi: 10.1186/s12906-018-2371-x. PMID 30453950